CLINICAL TRIAL: NCT04169906
Title: A Phase I Study of TS-142 in Non-Elderly Healthy Participants (Repeated Doses) (A Multiple Ascending Dose Study to Evaluate the Safety, Pharmacokinetics, and Pharmacodynamics of TS-142 in Non-Elderly Participants)
Brief Title: A Phase I Study of TS-142 in Healthy Participants (Repeated Doses)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taisho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: TS142-102
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2019-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — TS-142

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: TS-142, 10 mg; Drug: TS-142, 20 mg; Drug: TS-142, 30 mg
- TS-142 10 mg (Experimental)
  Interventions: Drug: Placebo; Drug: TS-142, 10 mg; Drug: TS-142, 20 mg; Drug: TS-142, 30 mg
- TS-142 20 mg (Experimental)
  Interventions: Drug: Placebo; Drug: TS-142, 10 mg; Drug: TS-142, 20 mg; Drug: TS-142, 30 mg
- TS-142 30 mg (Experimental)
  Interventions: Drug: Placebo; Drug: TS-142, 10 mg; Drug: TS-142, 20 mg; Drug: TS-142, 30 mg

INTERVENTIONS:
Drug: Placebo — Participants will receive placebo once daily for 7 consective days
Drug: TS-142, 10 mg — Participants will receive 10 mg of TS-142 once daily for 7 consective days
Drug: TS-142, 20 mg — Participants will receive 20 mg of TS-142 once daily for 7 consective days
Drug: TS-142, 30 mg — Participants will receive 30 mg of TS-142 once daily for 7 consective days

SUMMARY:
The purpose of this study is to investigate the safety, pharmacokinetics, and pharmacodynamics of repeated dosing of TS-142 when administered once daily to healthy Japanese non-elderly participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) ≥18.5 and <25.0 kg/m^2 at screening inspection

Exclusion Criteria:

* History of clinically relevant disease of some organ systems that may be considerd inappropriately for this study
* History of drug and food allergy

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2016-10-08 (Actual); Study Completion 2016-10-08 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-emergent Adverse Events (TEAEs) and Serious AEs (SAEs) | Day 1 up to Day 14
  Number of Treatment-emergent Adverse Events (TEAEs) and Serious AEs (SAEs) reported as mild, moderate, severe
Area under the concentration-time curve AUC (tau) | Day 1 up to Day 9
  Concentration of TS-142 and its metabolites in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Shigeru Okuyama, Study Director — Taisho Pharmaceutical Co., Ltd.
Locations (1):
- The medical facility selected by Taisho Pharmaceutical Co., Ltd, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kambe D, Hasegawa S, Imadera Y, Mano Y, Matsushita I, Konno Y, Ogo H, Uchimura N, Uchiyama M. Pharmacokinetics, pharmacodynamics and safety profile of the dual orexin receptor antagonist vornorexant/TS-142 in healthy Japanese participants following single/multiple dosing: Randomized, double-blind, placebo-controlled phase-1 studies. Basic Clin Pharmacol Toxicol. 2023 Nov;133(5):576-591. doi: 10.1111/bcpt.13930. Epub 2023 Sep 10. PMID 37563858